CLINICAL TRIAL: NCT03631433
Title: An Evaluation of Postoperative Pain Using Ibuprofen Versus Ibuprofen/Acetaminophen in Patients With Symptomatic Irreversible Pulpitis and Symptomatic Apical Periodontitis
Brief Title: Ibuprofen Versus Ibuprofen/Acetaminophen Postoperatively in Patients Needing Root Canal Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015H0433
Record Dates: First submitted 2018-08-09; First posted 2018-08-15 (Actual); Results first posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: identical appearing tablets and random allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ibuprofen (Active Comparator): A registered pharmacist compounded identical appearing tablets of 200 mg ibuprofen and tablets of 200 mg ibuprofen/216.7 mg acetaminophen. The tablets were placed in identical-appearing bottles (60 tabs of 200 mg ibuprofen or 60 tabs of a combination of 200 mg ibuprofen/216.7 mg acetaminophen). At the end of the debridement appointment, the patient received either a bottle containing 60 tabs of 200 mg ibuprofen or 60 tabs of 200 mg ibuprofen/216.7 mg acetaminophen. The patients were instructed to take 3 tablets every 6 hours as needed for pain.
  Interventions: Drug: Ibuprofen 600 mg
- ibuprofen/acetaminophen combination (Experimental): A registered pharmacist compounded identical appearing tablets of 200 mg ibuprofen and tablets of 200 mg ibuprofen/216.7 mg acetaminophen. The tablets were placed in identical-appearing bottles (60 tabs of 200 mg ibuprofen or 60 tabs of a combination of 200 mg ibuprofen/216.7 mg acetaminophen). At the end of the debridement appointment, the patient received either a bottle containing 60 tabs of 200 mg ibuprofen or 60 tabs of 200 mg ibuprofen/216.7 mg acetaminophen. The patients were instructed to take 3 tablets every 6 hours as needed for pain.
  Interventions: Drug: ibuprofen 600 mg and acetaminophen 650 mg

INTERVENTIONS:
Drug: Ibuprofen 600 mg — identical appearing tablets containing 600 mg of ibuprofen
  Arms: ibuprofen
Drug: ibuprofen 600 mg and acetaminophen 650 mg — identical appearing tablets of the combination of ibuprofen and acetaminophen
  Arms: ibuprofen/acetaminophen combination

SUMMARY:
Aim: The purpose of this study was to compare ibuprofen versus an ibuprofen/acetaminophen combination for postoperative pain control in patients requiring root canal treatment with a tooth that is painful to cold and biting.

Methodology: Following regular root canal treatment, patients randomly received identical appearing tablets of 600 mg ibuprofen or 600 mg ibuprofen/650 mg acetaminophen to be taken every 6 hours as needed for pain. A 4-day diary was used to record pain and medication use.

DETAILED DESCRIPTION:
This was a single-center, double-blind, interventional trial where (randomly) one group received ibuprofen and the other group received ibuprofen and acetaminophen.

Before the experiment, the ibuprofen and ibuprofen/acetaminophen groups were assigned 6-digit random numbers. The number assignment determined which drug regimen would be administered postoperatively for each patient. Only the random numbers were recorded on the data collection sheet in order to maintain blinding of the experiment.

The blinding of the ibuprofen and ibuprofen/acetaminophen medications was done as follows. A registered pharmacist compounded identical appearing tablets of 200 mg ibuprofen and tablets of 200 mg ibuprofen/216.7 mg acetaminophen. The tablets were placed in identical-appearing bottles (60 tabs of 200 mg ibuprofen or 60 tabs of a combination of 200 mg ibuprofen/216.7 mg acetaminophen). The pharmacist prepared the master code sheet and assigned the random numbers to the bottles. Therefore, the medication was blind to both the patient and the operator. A copy of the master list of random numbers was supplied by the compounding pharmacist solely to the lead researcher and was not made available to anyone else during the data collection period.

At the end of the debridement appointment, the patient received either a bottle containing 60 tabs of 200 mg ibuprofen or 60 tabs of 200 mg ibuprofen/216.7 mg acetaminophen. The patients were instructed to take 3 tablets every 6 hours as needed for pain.

The patients received a diary for 4 days post-treatment to record pain, percussion pain, and the amount and type of study medications taken. Patients were instructed to tap on the tooth that had emergency endodontic treatment and record this as their percussion pain. Patients recorded their pain levels on a VAS as described earlier for postoperative treatment pain. Starting on the morning after their appointment, patients also recorded the number of study medications taken within each 24-hour period.

ELIGIBILITY:
Inclusion Criteria:

1. mandibular (bottom) or maxillary (top) posterior (back) tooth requiring root canal treatment
2. mandibular (bottom) or maxillary (top) posterior (back) tooth with symptomatic irreversible pulpitis and symptomatic apical periodontitis (painful tooth to cold and biting)

2. between the ages of 18 and 65 years of age 3. American Society of Anesthesiologist classification I

Exclusion Criteria:

1. patients younger than 18 or older than 65 years of age
2. American Society of Anesthesiologist classification II or higher
3. allergies or contraindications to ibuprofen
4. allergies or contraindications to acetaminophen
5. pregnancy
6. inability to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-07-17 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ibuprofen | Ibuprofen/Acetaminophen Combination
Started | 49 | 53
Completed | 49 | 53
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ibuprofen/Acetaminophen: A registered pharmacist compounded identical appearing tablets of 200 mg ibuprofen and tablets of 200 mg ibuprofen/216.7 mg acetaminophen. The tablets were placed in identical-appearing bottles (60 tabs of 200 mg ibuprofen or 60 tabs of a combination of 200 mg ibuprofen/216.7 mg acetaminophen). At the end of the debridement appointment, the patient received either a bottle containing 60 tabs of 200 mg ibuprofen or 60 tabs of 200 mg ibuprofen/216.7 mg acetaminophen. The patients were instructed to take 3 tablets every 6 hours as needed for pain.
  ibuprofen 600 mg and acetaminophen 650 mg: identical appearing tablets of the combination of ibuprofen and acetaminophen
- Total: Total of all reporting groups
Arm/Group | Ibuprofen | Ibuprofen/Acetaminophen | Total
Number analyzed (Participants) | 49 | 53 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 53 | 102
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (11) | 35 (12) | 34 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 39 | 68
  Male | 20 | 14 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49 | 53 | 102
pain level on a Heft-Parker VAS [Mean (Standard Deviation); unit: units on a scale] | 129 (22) | 128 (23) | 128 (22)

OUTCOME MEASURES:

1. Primary Outcome: Heft Parker Visual Analog Scale Pain Scale Pain Measurements
Description: Heft-Parker Visual Analog Scale measurements (0-170mm scale) Higher values are a worse outcome.
Time Frame: 4 day postoperative survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ibuprofen | Ibuprofen/Acetaminophen Combination
Number analyzed (Participants) | 49 | 53
units on a scale | 63 (41) | 60 (42)

2. Primary Outcome: Number of Participants
Description: Number of participants requiring escape pills
Time Frame: 4 day postoperative survey
Measure: Count of Participants; unit: Participants
Arm/Group | Ibuprofen | Ibuprofen/Acetaminophen Combination
Number analyzed (Participants) | 49 | 53
Participants | 20 | 18

ADVERSE EVENTS:
Time Frame: Throughout the study - approximately 1 year
Description: This was a low risk study, patients medically healthy (ASA I) taking over the counter medication for it's approved purpose.
  All-Cause Mortality and Serious Adverse Events were not monitored/assessed.
Arm/Group | Ibuprofen | Ibuprofen/Acetaminophen Combination
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/49 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT03631433/Prot_SAP_000.pdf